CLINICAL TRIAL: NCT04833530
Title: The Effect of Preoperative Anxiety, Extent of Ovarian Stimulation, and Positive Pressure Ventilation on Gastric Antrum Size in Women Undergoing Oocyte Pickup for in Vitro Fertilization Under General Anaesthesia.
Brief Title: The Effect of Preoperative Anxiety, on Gastric Antrum Size in Women Undergoing in Vitro Fertilization
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0010-21
Record Dates: First submitted 2021-03-20; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Woman undergoing an gastric ultrasound assessment.: Woman undergoing general anesthesia for oocyte retrieval during in vitro fertilization, will undergo an gastric ultrasound assessment.
  Interventions: Diagnostic Test: Gastric Ultrasound

INTERVENTIONS:
Diagnostic Test: Gastric Ultrasound — In the operating room, a gastric ultrasound will be performed in the supine position and the antral cross sectional area will be measured. Anesthesia will be induced in standard procedure and positive pressure will be instituted according to the standard protocol accepted in our hospital.
  At the end of the procedure, the gastric ultrasound circumference will be measured again.

SUMMARY:
Pulmonary aspiration is one of the most serious risks of general anesthesia and has been reported to occur in as many as 1 in 4000 cases of general anesthesia. Gastric ultrasound is an emerging point-of-care tool that provides bedside information on gastric content and volume.

There have been a few factors which are thought to increase gastric size. Delayed gastric emptying such as caused by gastroparesis in Diabetes Mellitus is an example. Certain surgeries also cause gastroparesis. Other preoperative factors including pain, preoperative anxiety, and blood levels of estradiol or progesterone are less well studied.

DETAILED DESCRIPTION:
Women will be recruited before undergoing the procedure.

Upon signed informed consent, women will be asked to rank their anxiety level on a scale of 0-10 (Verbal Numeric Anxiety Score). This scale has been used for previous studies to assess anxiety (Orbach-Zinger, Danon)

In the operating room, a gastric ultrasound will be performed in the supine position and the antral cross sectional area will be measured. This study is purely observational, the gastric ultrasound assessment is non-invasive and will not cause any adverse effects or discomfort to the patient. Participation in the study will not affect clinical management in any way.

Each one of the ultrasound assessments will be performed by one of the study's' investigators.

Anesthesia will be induced in standard procedure and positive pressure will be instituted according to the standard protocol accepted in our hospital.

At the end of the procedure, the gastric ultrasound circumference will be measured again.

ELIGIBILITY:
Inclusion Criteria:

Woman aged 18 and above undergoing general anesthesia for oocyte retrieval during in vitro fertilization with the ability to sign an informed consent.

Exclusion Criteria:

1. Women with BMI >40
2. Women with diabetes
3. Women who have previously undergone gastric surgery
4. Women with language barriers.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman aged 18 and above undergoing general anesthesia for oocyte retrieval during in vitro fertilization with the ability to sign an informed consent.
Study Population: Woman aged 18 and above undergoing general anesthesia for oocyte retrieval during in vitro fertilization with the ability to sign an informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative gastric ultrasound measurement | Within 24 hours before Oocyte pickup
Post-anesthesia gastric ultrasound measurement | During Oocyte pickup 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Orbach-zinger, Principal Investigator — Rabin Medical Center
Locations (1):
- Beilinson hospital, Petach Tikvah, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Azem K, Orbach-Zinger S, Heesen P, Finkelstein A, Eidelman LA, Shufaro Y, Arzola C. The effect of preoperative anxiety and ovarian stimulation on gastric antrum size: a prospective observational study. J Psychosom Obstet Gynaecol. 2023 Dec;44(1):2170226. doi: 10.1080/0167482X.2023.2170226. PMID 36774546